CLINICAL TRIAL: NCT05958576
Title: Effect of Age on Sperm Recovery of Microdissection Testicular Sperm Extraction in Nonobstructive Azoospermia Patients
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 78070
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-12

CONDITIONS: Non-obstructive Azoospermia
Keywords: non-obstructive azoospermia; microdissection testicular sperm extraction; sperm retrieval rate; age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Males with non-obstructive azoospermia (NOA) have an opportunity to obtain sperm by treatment with microdissection testicular sperm extraction (mTESE), gold-standard surgical technique for them. The overall sperm retrieval rate (SRR) of mTESE in NOA patients is about 50%, but the predictive factors of SRR remain were understudied, especially the effect of age. The purpose of this study was to explore the factors influencing the SRR of mTESE in NOA patients with different etiologies.

Methods: This observational study recruit NOA patients treated with their first mTESE. The stratified research was used to investigate SRR by dividing patients into seven groups based on etiology. The primary outcome was SRR. Multivariable logistic regression was used to analyze the factors influencing SRR.

DETAILED DESCRIPTION:
As the most severe form of infertility, azoospermia is observed in approximately 10% to 15% of infertile males and can be classified as obstructive azoospermia (OA) and non-obstructive azoospermia (NOA), the latter of which cause spermatogenic dysfunction. Approximately 60% of NOA males are diagnosed with congenital, acquired, or idiopathic NOA (iNOA). The most common congenital causes of NOA are Klinefelter syndrome (KS) and Y chromosome azoospermia factor (AZF) deletions, whereas the acquired causes of NOA are mumps orchitis, cryptorchidism, cryptozoospermia, and iatrogenic causes (chemotherapy, radiotherapy, hypogonadotropic hypogonadism). For iNOA, the most common form of NOA, there is no clear cause in approximately 50-80% of cases.

As a prevalent chromosomal abnormality, KS with two or more X chromosomes is the most common form of congenital NOA that affects approximately 3-4% of infertile males and more than 10% of azoospermic males. The incidence of Y-chromosome AZF microdeletions in fertile males is 0.025%, but it increases to 2%-10% in infertile males. Mumps orchitis is the most common and serious complication of mumps virus infection in adolescents and young adults, with an incidence of 40% in males with postpubertal mumps, and approximately 30% of males suffer from infertility or subfertility. As an extremely severe form of oligozoospermia, cryptozoospermia is characterized by the absence of sperm in semen by microscopic examination but the presence of sperm in centrifuge sediment, with an incidence of approximately 8.73% in infertile males. Cryptorchidism represents one of the most common urogenital abnormalities in childhood, affecting 1.1%-45% of preterm and 1%-4.6% of full-term infants, and approximately 10% of infertile males have a history of cryptorchidism.

Obtaining sperm by microdissection testicular sperm extraction (mTESE) is the primary treatment approach for males with NOA. The average sperm retrieval rate (SRR) in NOA males is approximately 50%, however, NOA patients with different etiologies have different SSRs ranging from 30% to 75%, with the highest and lowest SRRs corresponding to those with a history of mumps orchitis and iNOA, respectively. The predictive factors of SRR in males with NOA treated with mTESE include age; testis volume; serum follicle stimulating hormone (FSH), testosterone (T), inhibin B, and anti-Müllerian hormone (AMH) levels and testicular histopathology. However, the relationship between SSR and age in NOA patients undergoing mTESE is unclear, with several studies reporting no association between SSR and age or a negative correlation between SSR and age. Other studies have reported that older age was predictive of successful sperm retrieval.

The goal of this study was to analyze the factors influencing the SRR in NOA patients with different etiologies treated with mTESE based on age, body mass index (BMI), testis volume hormone levels and infertility duration in a large cohort. Our findings provide valuable information on the likelihood of successful mTESE. Therefore, preoperative evaluations based on the information provided in this study will help patients and surgeons in selecting the best approach by shared decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Non-obstructive azoospermia patients were treated with microdissection testicular sperm extraction.

Exclusion Criteria:

* Obstructive azoospermia patients.
* Fertile males.

Ages: 21 Years to 57 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Non-obstructive azoospermia patients
Sampling Method: Non-Probability Sample
Enrollment: 3104 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
sperm retrieval rate | immediately after surgery
  If sperm was observed during the surgery, this case was defined as positive. If sperm wasn't observed, the case was defined as negative.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Ph.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD of this study is openly available to other researchers. You could get them from Li Zhang and please contact her (lizhang0814@163.com).

REFERENCES:
- [Result] Mittal PK, Little B, Harri PA, Miller FH, Alexander LF, Kalb B, Camacho JC, Master V, Hartman M, Moreno CC. Role of Imaging in the Evaluation of Male Infertility. Radiographics. 2017 May-Jun;37(3):837-854. doi: 10.1148/rg.2017160125. Epub 2017 Apr 14. PMID 28410062
- [Result] Tuttelmann F, Werny F, Cooper TG, Kliesch S, Simoni M, Nieschlag E. Clinical experience with azoospermia: aetiology and chances for spermatozoa detection upon biopsy. Int J Androl. 2011 Aug;34(4):291-8. doi: 10.1111/j.1365-2605.2010.01087.x. Epub 2010 Jun 28. PMID 20609027
- [Result] Hopps CV, Mielnik A, Goldstein M, Palermo GD, Rosenwaks Z, Schlegel PN. Detection of sperm in men with Y chromosome microdeletions of the AZFa, AZFb and AZFc regions. Hum Reprod. 2003 Aug;18(8):1660-5. doi: 10.1093/humrep/deg348. PMID 12871878
- [Result] Forti G, Corona G, Vignozzi L, Krausz C, Maggi M. Klinefelter's syndrome: a clinical and therapeutical update. Sex Dev. 2010 Sep;4(4-5):249-58. doi: 10.1159/000316604. Epub 2010 Jul 21. PMID 20664188
- [Result] Krausz C. Male infertility: pathogenesis and clinical diagnosis. Best Pract Res Clin Endocrinol Metab. 2011 Apr;25(2):271-85. doi: 10.1016/j.beem.2010.08.006. PMID 21397198
- [Result] Pena VN, Kohn TP, Herati AS. Genetic mutations contributing to non-obstructive azoospermia. Best Pract Res Clin Endocrinol Metab. 2020 Dec;34(6):101479. doi: 10.1016/j.beem.2020.101479. Epub 2020 Dec 15. PMID 33390350
- [Result] Ternavasio-de la Vega HG, Boronat M, Ojeda A, Garcia-Delgado Y, Angel-Moreno A, Carranza-Rodriguez C, Bellini R, Frances A, Novoa FJ, Perez-Arellano JL. Mumps orchitis in the post-vaccine era (1967-2009): a single-center series of 67 patients and review of clinical outcome and trends. Medicine (Baltimore). 2010 Mar;89(2):96-116. doi: 10.1097/MD.0b013e3181d63191. PMID 20517181
- [Result] Mieusset R, Bujan L, Massat G, Mansat A, Pontonnier F. Clinical and biological characteristics of infertile men with a history of cryptorchidism. Hum Reprod. 1995 Mar;10(3):613-9. doi: 10.1093/oxfordjournals.humrep.a135998. PMID 7782441
- [Result] Zhang HL, Zhao LM, Mao JM, Liu DF, Tang WH, Lin HC, Zhang L, Lian Y, Hong K, Jiang H. Sperm retrieval rates and clinical outcomes for patients with different causes of azoospermia who undergo microdissection testicular sperm extraction-intracytoplasmic sperm injection. Asian J Androl. 2021 Jan-Feb;23(1):59-63. doi: 10.4103/aja.aja_12_20. PMID 32341210
- [Result] Bonarriba CR, Burgues JP, Vidana V, Ruiz X, Piza P. Predictive factors of successful sperm retrieval in azoospermia. Actas Urol Esp. 2013 May;37(5):266-72. doi: 10.1016/j.acuro.2012.06.002. Epub 2012 Oct 9. English, Spanish. PMID 23062736